CLINICAL TRIAL: NCT03822962
Title: Post-operative Pain Management Following Functional Endoscopic Sinus Surgery
Brief Title: Pain Management Following Sinus Surgery
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Decrease in accrual during the COVID-19 pandemic and several sites withdrawing
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0417-18-FB
Record Dates: First submitted 2019-01-28; First posted 2019-01-30 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Nasal Sinus; Inflammation; Opioid Abuse; Pain, Postoperative
Keywords: NSAIDs; post-operative pain; post-operative hemorrhage; Functional endoscopic sinus surgery
MeSH Terms: conditions — Sinusitis; Opioid-Related Disorders; Pain, Postoperative; Postoperative Hemorrhage | interventions — Ibuprofen; Tablets; Acetaminophen

STUDY DESIGN:
Intervention Model Description: prospective, cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard Tylenol Regimen (Other): Patient will be given a standard regimen:
  Tylenol 1000 mg by mouth every 6 hours scheduled and a rescue prescription of oxycodone 5 mg tablets by mouth every 6 hours as needed for pain. Ten total oxycodone tablets will be prescribed.
  Interventions: Other: Standard Regimen | Tylenol
- Ibuprofen 600mg (Active Comparator): Tylenol 1000 mg by mouth every 6 hours scheduled and ibuprofen 600 mg tablet by mouth every 8 hours scheduled and a rescue prescription of oxycodone 5 mg tablets by mouth every 6 hours as needed for pain. Ten total oxycodone tablets will be prescribed.
  Interventions: Drug: Ibuprofen 600Mg Tablet; Other: Standard Regimen | Tylenol

INTERVENTIONS:
Drug: Ibuprofen 600Mg Tablet — ibuprofen 600 mg by mouth every 8 hours scheduled in addition to standard tylenol regimen.
  Other Names: Advil, Motrin IB
  Arms: Ibuprofen 600mg
Other: Standard Regimen | Tylenol — Tylenol 1000 mg by mouth every 6 hours scheduled and a rescue prescription of oxycodone 5 mg tablets by mouth every 6 hours as needed for pain. Ten total oxycodone tablets will be prescribed.
  Other Names: Acetaminophen

SUMMARY:
This Study evaluates the effect of adding Non-steroidal anti-inflammatories (NSAIDs) to the post-operative pain management of sinus surgery patients and wether or not this addition reduces or eliminates the need for narcotic pain medications.

Patients will be instructed to take an NSAID regimen after surgery and will be instructed to take narcotics only for breakthrough pain.

DETAILED DESCRIPTION:
National attention has been given to the concerning rise of opioid abuse in this country, with prescriptions for this medications more than quadrupaling in the last 17 years.

Little is known as to the appropriate use of opioid analgesics in the post-operative recovery of patients undergoing sinus surgery. Furthermore, most pain protocols include only Tylenol based opioid analgesics. No study has prospectively evaluated the volume of use of Tylenol based opioid analgesics and whether the addition of NSAIDS decreased the need for opioid analgesics.

This study will compare opioid use with and without the addition of NSAIDS following sinus surgery.

Post-operative opioid use is a great public health concern, relatively unstudied, and an area with an opportunity for potential intervention to significantly reduce risks, morbidity, and mortality to our postoperative patients by better formulating a postoperative pain management plan using evidence-based practices. Appropriate opioid prescribing practices can reduce the risk of addiction, drug overdose, death, and undertreated pain. By optimizing post-operative pain management protocols, the need for opioids following sinus surgery should be minimized.

ELIGIBILITY:
Inclusion Criteria:

• All patients age 18-65 undergoing functional endoscopic sinus surgery +/- nasal airway surgery (septoplasty and/or inferior turbinate reduction).

Exclusion Criteria:

* Not taking anti-coagulation medications including aspirin
* Clinical Diagnosis of aspirin-exacerbated respiratory disease
* Clinical Diagnosis of Cystic Fibrosis
* Clinical Diagnosis of Primary Ciliary Dyskinesia
* Inclusion of a Draf III frontal sinusotomy
* Clinical Diagnosis of Liver/Kidney Failure
* Clinical Diagnosis of Thrombocytopenia
* Clinical Diagnosis of Poorly controlled hypertension
* Clinical Diagnosis of Recent GI ulcers or gastritis
* Clinical Diagnosis of Chronic pain as defined by a narcotic prescription with 6 months or involvement in a pain management program
* Clinical Diagnosis of Primary Headache disorder
* The use of nasal decongestants in the post-operative period.
* The use of nasal packing or absorbable biomaterials.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-11-07 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Pain level | 1 week
  Patients will be given a Visual Analogue scale to help document their level of pain from Post-operative days 0, 1, 2, 3, 4 ,5 and the first post-operative visit with the surgeon. The patient will measure their pain score each time they take medication.
  The pain scale called the Wong-Baker FACES pain rating scale is a 0-10 pain scale. 0 = no hurt, 2 = hurts little bit, 4 = hurts little more, 6 = hurts even more, 8 = hurts whole lot, 10 = hurts worst. The numbers are added up to a sum and put into their perspective category known by the Otolaryngologist.

SECONDARY OUTCOMES:
Rate of bleeding | 1 week
  Any physician visits secondary to bleeding will be tabulated including ER and office visits.

CONTACTS AND LOCATIONS:
Overall Officials: Christie Barnes, MD, Principal Investigator — University of Nebraska
Locations (2):
- United States (2):
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University of Cincinnati, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No